CLINICAL TRIAL: NCT04632693
Title: Soft Tissue Augmentation Using Coronally Advanced Flap With Either Subepithelial Connective Tissue and Vitamin C Versus Subepithelial Connective Tissue Graft Alone in Management of RT1 Gingival Recession
Brief Title: Soft Tissue Augmentation Using CAF With Either SCTG and Vitamin C Versus SCTG Alone in Management of RT1 Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Andrew Albert Anwar Zaki, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-6-20
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Gingival Thickness
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF with SCTG and vitamin C (Experimental): Coronally advanced flap with subepithelial connective tissue graft and vitamin C.
  Interventions: Procedure: CAF with SCTG and Vitamin C injection
- CAF with SCTG (Active Comparator): Coronally advanced flap with subepithelial connective tissue graft.
  Interventions: Procedure: CAF with SCTG alone

INTERVENTIONS:
Procedure: CAF with SCTG and Vitamin C injection — Injection of vitamin C after CAF with SCTG aiming to increase gingival thickness in patients with RT1 gingival recession.
  Arms: CAF with SCTG and vitamin C
Procedure: CAF with SCTG alone — Coronally advanced flap with subepithelial connective tissue graft.
  Arms: CAF with SCTG

SUMMARY:
Compare gingival thickness following CAF With SCTG and Vitamin C Versus SCTG Alone in Management of RT1 Gingival Recession.

DETAILED DESCRIPTION:
Control group (coronally advanced flap and subepithelial connective tissue graft alone) Test group (coronally advanced flap and subepithelial connective tissue graft using microsurgical approach) Same procedure will be executed but with the addition of vitamin C injection. Intraepidermal injection (oral mesotherapy technique) of 1-1.5 ml (200-300 mg concentration) of L-ascorbic acid will be done. It will be locally introduced in relation to the keratinized gingival tissues with extension to the whole target region successively using special syringes (30 gauge). The needle will be introduced parallel to the gingival tissues with the bevel facing upwards. Vitamin C will then be delivered through the attached gingival tissues at the epithelium-connective tissue junction (equivalent to epidermal- dermal junction) till the tissues blanch. Vitamin C will be injected first time immediately postsurgical and then repeated once per week for 3 consecutive weeks for a total of 4 injections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older.
2. Periodontally and systemically healthy.
3. Buccal recession defects classified as Cairo RT1.
4. Presence of identifiable CEJ (Zucchelli et al., 2010).
5. Clinical indication and/or patient request for recession coverage.
6. O'Leary index less than 20% (O'Leary, Drake and Naylor, 1972).

Exclusion Criteria:

1. Cairo RT2 or RT3 recession defects.
2. Pregnant females.
3. Smokers as smoking is a contraindication for any periodontal plastic surgery (Khuller, 2009).
4. Handicapped and mentally retarded patients.
5. Patients undergoing radiotherapy.
6. Teeth with cervical restorations, abrasion and malalignment.
7. Presence of systemic disease that would affect wound healing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Ginigval thickness | 6 months
  Determined 2 mm apical to the gingival margin with a short needle for anesthesia and a 3 mm diameter silicon disk stop. The needle is inserted perpendicular to the mucosal surface, through the soft tissues with light pressure until a hard surface is felt. The silicon disk stop is then placed in tight contact with the soft tissue surface with the coronal border overlapping the soft tissue margin. As the needle is located in the center of the silicon disk, measurement of GT is performed 2 mm apical from the gingival margin. Once in the correct position, the disk is fixed with a drop of cyanocrylic adhesive; after careful removal of the needle, the penetration depth is measured with a caliper accurate to the nearest 0.1 mm.

SECONDARY OUTCOMES:
Root Coverage Esthetic Score | 6 months
  A system proposed for evaluating esthetic outcomes of root coverage procedures. The RES system evaluated five variables at 6-months after surgery: the level of the gingival margin, marginal tissue contour, soft tissue texture, MGJ alignment, and gingival color.
Early Healing Index | 6 months
  A system proposed for the clinical assessment of the early wound events by using a differentiated early wound healing index (EHI) (Wachtel et al., 2003).
Gingival Recession Depth (RD) | 6 months
  Measured from the CEJ to the most apical extension of the gingival margin.
Gingival Recession Width (RW) | 6 months
  Measured horizontally between the borders of the recession at the level of CEJ.
Percentage of root coverage | 6 months
  (Preoperative vertical recession - Postoperative vertical recession/preoperative vertical recession) x 100.
Probing Depth (PD) | 6 months
  Measured from the gingival margin to the bottom of the gingival sulcus.
Clinical Attachment Level (CAL) | 6 months
  Measured from the CEJ to the bottom of the gingival sulcus.
Height of Keratinized Tissue (KTH) | 6 months
  Measured as the distance between the gingival margin and the mucogingival junction (MGJ).
  All measurements will be performed by means of the UNC periodontal probe and will be rounded up to the nearest millimeter.
Post-Operative Pain | 2 weeks
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first 2 weeks postoperatively.
Post-Surgical Patient Satisfaction | 6 months
  A 3-item questionnaire is asked and the patients shall use a 7-point answer scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine - CU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided